CLINICAL TRIAL: NCT06117982
Title: Does Subcutaneous Granulocyte Colony Stimulating Factor (G-CSF) Improve Ovarian Reserve in Women With Premature Ovarian Insufficiency?
Brief Title: The Impact of Granulocyte Colony Stimulating Factor on Premature Ovarian Insufficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trio Fertility (Other)
Responsible Party: Principal Investigator, Dr. Robert F. Casper, Scientific Director, MD, FRCSC, REI, Trio Fertility
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TF005
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Primary Ovarian Insufficiency; Premature Ovarian Failure
Keywords: Filgrastim; Granulocyte colony stimulating factor; Premature Ovarian Insufficiency; Neupogen
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patients with POI receiving G-CSF injections (Experimental): Patients will receive 0.5 ml SC injections of G-CSF (Neupogen, Amgen, USA) at 300 micrograms/day for 4 consecutive days. The first injection will be administered in our office with a 60-minute observation period. Subsequent injections can be self-administered at home for three days, with a return to our clinic for monitoring the following day. This 4-day Neupogen regimen will be repeated in one month.
  Patients may undergo two rounds of G-CSF treatment one month apart. If no improvement is observed in gonadotropin, anti-Mullerian levels, and antral follicle count, a third treatment may be offered a month later. Follow-up includes blood assessment of AMH and FSH, as well as ultrasound measurement of basal antral follicle count for three months after the last G-CSF infusion.
  Interventions: Drug: Neupogen

INTERVENTIONS:
Drug: Neupogen — Subcutaneous injection of 0.5 ml of Neupogen at a concentration of 300 micrograms/day for 4 consecutive days
  Other Names: Filgrastim

SUMMARY:
The goal of this pilot study is to improve ovarian reserve markers in patients with premature ovarian insufficiency. The main question it aims to answer is:

- Will treatment with G-CSF allow improvement in markers of ovarian reserve?

DETAILED DESCRIPTION:
The research team hypothesize that treatment of premature ovarian insufficiency patients with G-CSF to mobilize bone marrow hematopoietic stem cells will allow for improved ovarian reserve markers including antral follicle count, anti-Mullerian hormone (AMH) levels and gonadotropin (FSH) levels. The research team anticipate these outcomes:

* Primary outcome: Decreased serum FSH and increased AMH levels and u/s measurement of increased antral follicle count (AFC)
* Secondary outcome: Improved ovarian response in IVF cycles if BAFs develop, and spontaneous or IVF pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 25-40
* Woman who meet criteria for POI defined as AFC < 5, AMH < 3 pmol/L and FSH >30 IU/L. There may also be associated symptoms of the menopause such as hot flushes, night sweats, insomnia and vaginal dryness.
* Women who are not taking any other medical or fertility treatments except natural estrogen to stop hot flushes.
* Those who are provided with informed consent.

Exclusion Criteria:

* Women with age > 40
* Women with history of autoimmune disorders
* Women with a history of hematopoietic cell malignancies
* Women with sickle cell disease
* Women with any other comorbidities that would preclude infertility treatment and pregnancy such as HIV/AIDS, hepatitis B or C, breast cancer or body mass index (BMI) >40.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Improving ovarian reserve markers | It is anticipated within six months
  Success of the treatment will be assessed by a change in serum FSH, AMH (measure of ovarian reserve) and number of antral follicles (AFC).

SECONDARY OUTCOMES:
Successful Pregnancy | It is anticipated after the first six months of the study time frame
  If a change in the number of basal antral follicles is seen in association with an FSH level below 20 IU/L, the subjects will be offered a cycle of IVF to see if oocytes and subsequently embryos can be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Robert F. Casper, Dr., Principal Investigator — Trio Fertility, Toronto, ON, Canada
Locations (1):
- Trio Fertility, Toronto, Ontario, Canada

REFERENCES:
- [Result] Hershlag A, Schuster MW. Return of fertility after autologous stem cell transplantation. Fertil Steril. 2002 Feb;77(2):419-21. doi: 10.1016/s0015-0282(01)02987-9. PMID 11821109
- [Result] Salooja N, Szydlo RM, Socie G, Rio B, Chatterjee R, Ljungman P, Van Lint MT, Powles R, Jackson G, Hinterberger-Fischer M, Kolb HJ, Apperley JF; Late Effects Working Party of the European Group for Blood and Marrow Transplantation. Pregnancy outcomes after peripheral blood or bone marrow transplantation: a retrospective survey. Lancet. 2001 Jul 28;358(9278):271-6. doi: 10.1016/s0140-6736(01)05482-4. PMID 11498213
- [Result] Pellicer, N, Herraiz, S, Romeu, M, Martinez, S, Buiges, A, Gomez-Seguí, I, Martínez, J, Pellicer, A., 2020. Bone marrow derived stem cells restore ovarian function and fertility in women with POI: Interim report of a randomized trial comparing mobilization versus ovarian injection. 36th Annual Meeting of European Society Reproduction and Embryology (ESHRE).
- [Derived] Sadeghi Y, Deda L, Albar M, Casper R. Granulocyte colony-stimulating factor treatment in women with premature ovarian insufficiency: a pilot clinical study of biological activity and menstrual resumption. Reprod Biol Endocrinol. 2026 Jan 7;24(1):19. doi: 10.1186/s12958-025-01510-z. PMID 41495818
- See also: Bone marrow derived stem cells restore ovarian function and fertility in premature ovarian insufficiency women. Interim report of a randomized trial: mobilization versus ovarian injection — http://www.ivi-rmainnovation.com/wp-content/uploads/2020/07/O-088-Bone-marrow-derived-stem-cells-restore-ovarian-function.pdf

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-07-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT06117982/Prot_ICF_000.pdf